CLINICAL TRIAL: NCT06772025
Title: Methodology Study in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass to Investigate Mechanisms Involved in Cardiac Surgery-associated Acute Kidney Injury.
Brief Title: A Study to Understand How Cardiac Surgery-associated Acute Kidney Injury Develops in Participants Who Undergo Heart Surgery With the Use of Heart-lung Machine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22785
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery-associated Acute Kidney Injury
Keywords: CSA-AKI; Cardiac surgery; Cardiopulmonary bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac surgery (Experimental): Patients scheduled for cardiac surgery with cardiopulmonary bypass will be managed according to local standard medical care. Blood and urine will be obtained pre-surgery and post-surgery for analysis.
  Interventions: Other: No investigational study intervention

INTERVENTIONS:
Other: No investigational study intervention — No investigational study interventions will be administered in this study. Participants will undergo therapeutic and diagnostic procedures as per local standard medical care and as deemed appropriate by the treating physicians. Collection of blood (not exceeding 200 mL) and urine samples and of available clinical data are the only activities performed in addition.

SUMMARY:
Researchers are looking for a better way to treat and prevent cardiac surgery-associated acute kidney injury (CSA-AKI) in people who undergo heart surgeries.

CSA-AKI is a common complication in people undergoing heart surgeries, where the kidneys stop working properly. CSA-AKI risk factors include older age and alongside diseases such as kidney disease and diabetes. Longer time with heart-lung machine during heart surgeries also increases the occurrence of CSA-AKI.

In this study, researchers want to better understand how CSA-AKI develops (also known as the mechanisms involved in the development of CSA-AKI) in people under heart surgeries, the presence of certain biomarkers in the body, especially with a focus on the early hours and days after the surgery. (A biomarker is a biological molecule found in blood, other body fluids, or tissues that is a sign of a normal or abnormal process, or of a condition or disease.) These biomarkers will be compared in participants who develop CSA-AKI within a week after heart surgery with the participants who do not develop CSA-AKI. The relationship with biomarkers will be determined by examining participants' blood and urine samples before and after surgery.

This may help researchers better understand CSA-AKI, identify potential treatment targets and develop possible treatments to prevent CSA-AKI.

Participants in this study will be people who have heart surgery already scheduled by their own doctors and have a risk of developing CSA-AKI. Participants will not receive any treatment as part of this study. They will undergo the heart surgery and related medical processes as per their normal medical treatment and management.

Each participant will be in the study for up to 2 months. During the study, the doctors and their study team will:

* collect participants' blood and urine samples before and after surgery
* assess participants' medical records and test reports during hospitalization
* monitor overall health of the participants throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of signing the informed consent form (ICF).
* Participants who are scheduled for hospital admission for any of the following cardiovascular surgery interventions, alone or in combination, involving cardiopulmonary bypass (CPB):

  * Aortic, mitral, or tricuspid valve surgery (repair or replacement)
  * Aortic surgery
  * ≥3 coronary artery bypass grafts
* Participant with: chronic kidney disease (CKD): 30 ≤ estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m^2

Exclusion Criteria:

* Emergency surgery situation
* Anemia - hemoglobin <10 g/dL
* Clinical signs of systemic infection or other infection requiring anti-infective treatment (viral, bacterial, fungal, parasitic; single-dose prophylaxis allowed)
* Systemic immunosuppressive or anti-inflammatory treatment including corticosteroids >10 mg prednisolone equivalent/day
* Any anti-cancer treatment within 3 months (e.g. immunotherapy, chemotherapy, radiotherapy)
* Major surgery within 2 months
* AKI within the last month
* Prior renal transplants or RRT
* Planned use of contrast media within 5 days prior to surgery or during surgery
* Patient included in an interventional clinical trial involving a pharmacological intervention
* Any reason that would make participation unadvisable, at the discretion of the investigator.
* Autoimmune disorders such as anti-glomerular basement membrane (anti-GBM) diseases, systemic lupus erythematosus, chronic rheumatic heart diseases, acute rheumatic heart pericarditis, endocarditis, myocarditis, rheumatic mitral valve diseases, rheumatic aortic valve diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with CSA-AKI until Day 3 post-surgery | Up to 3 days post surgery
  CSA-AKI: cardiac surgery-associated acute kidney injury

SECONDARY OUTCOMES:
Observed values of pre-defined biomarkers overall and by CSA-AKI outcome | Up to 7 days post surgery
  Non-genetic biomarkers will be investigated from blood, plasma, and urine collected in this study. CSA-AKI: cardiac surgery-associated acute kidney injury
Change from baseline of pre-defined biomarkers overall and by CSA-AKI outcome | Up to 7 days post surgery
  Non-genetic biomarkers will be investigated from blood, plasma, and urine collected in this study. CSA-AKI: cardiac surgery-associated acute kidney injury
Ratio to baseline of pre-defined biomarkers overall and by CSA-AKI outcome | Up to 7 days post surgery
  Non-genetic biomarkers will be investigated from blood, plasma, and urine collected in this study. CSA-AKI: cardiac surgery-associated acute kidney injury

CONTACTS AND LOCATIONS:
Locations (4):
- Herz- und Diabeteszentrum Nordrhein-Westfalen (HDZ NRW), Bad Oeynhausen, North Rhine-Westphalia, Germany
- United Kingdom (3):
  - Royal Papworth Hospital NHS Foundation Trust | Royal Papworth Hospital - Cardiac Surgery, Cambridge, Cambridgeshire
  - Guy's and St Thomas' NHS Foundation Trust | Harefield Hospital - Cardiology, Harefield, Greater London
  - Guy's and St Thomas' NHS Foundation Trust | Guy's & St Thomas' Hospital - Department of Critical Care & Nephrology, London, Greater London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22785